CLINICAL TRIAL: NCT01052350
Title: Investigations of Dementia in Parkinson Disease
Brief Title: PET Imaging in Parkinson Disease Dementia
Status: Active, not recruiting | Type: Observational
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: 06-0706-201103106
Record Dates: First submitted 2010-01-15; First posted 2010-01-20 (Estimated); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Parkinson's Disease
Keywords: Parkinson disease; PET imaging; PIB; dementia
MeSH Terms: conditions — Parkinson Disease; Dementia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood
Oversight: Data Monitoring Committee: No | US Export: No

GROUPS / COHORTS (2):
- Parkinson disease: individuals with Parkinson disease
- healthy control: individuals without Parkinson disease

SUMMARY:
The purpose of this study is to use a brain imaging method called PIB PET to determine dementia subtypes in patients with Parkinson's disease. The ultimate goal of this project is to be able to identify individuals with PD who are at risk of developing dementia, and to distinguish the underlying cause of dementia.

DETAILED DESCRIPTION:
The purpose of this study is to use a brain imaging method called PIB PET to determine dementia subtypes in patients with Parkinson's disease. The ultimate goal of this project is to be able to identify individuals with PD who are at risk of developing dementia, and to distinguish the underlying cause of dementia. We will be including both PD and normal subjects in this study. This a long term study and we are considering including a total of 320 participants in this protocol.

ELIGIBILITY:
Inclusion Criteria:

* PD patients must exhibit three of the following cardinal signs: rest tremor, rigidity, bradykinesia, or postural instability; or two of these features with one of the first three displaying asymmetry.

Exclusion Criteria:

* history of head trauma, major neurological or psychiatric diseases other than Parkinson disease and dementia, e.g. stroke, multiple sclerosis, depression or schizophrenia
* severe systemic diseases
* inability to lie still for 90 minutes
* metallic implants, pacemakers, or any other contraindication to MRI
* refusal to consent to brain donation

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants with and without Parkinson disease will be recruited from the Movement Disorders Center at Washington University, the St. Louis metro area, and throughout the midwest region.
Sampling Method: Non-Probability Sample
Enrollment: 320 (Estimated)
Dates: Start 2006-08; Primary Completion 2030-07 (Estimated); Study Completion 2030-07 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Joel S. Perlmutter, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- NeuroClinical Research Unit (NCRU), Washington University School of Medicine, St Louis, Missouri, United States